CLINICAL TRIAL: NCT00609622
Title: A Randomized, Phase 2B Study Of Sunitinib Plus Oxaliplatin, 5-Fluorouracil And Leucovorin (FOLFOX) Versus Bevacizumab Plus FOLFOX As First-Line Treatment In Patients With Metastatic Colorectal Cancer
Brief Title: Randomized Study Of Sunitinib Plus FOLFOX Versus Bevacizumab Plus FOLFOX In Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181104
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Neoplasms
Keywords: metastatic colorectal cancer sunitinib (Sutent) bevacizumab (Avastin) randomized study
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sunitinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Treatment arm A - sunitinib plus mFOLFOX6
  Interventions: Drug: sunitinib; Drug: mFOLFOX6
- B (Active Comparator): Treatment arm B - bevacizumab plus mFOLFOX6
  Interventions: Drug: bevacizumab; Drug: mFOLFOX6

INTERVENTIONS:
Drug: sunitinib — Sunitinib: 37.5 mg/day, oral, administered on an outpatient basis for 4 weeks on, 2 weeks off (Schedule 4/2).
  Other Names: Sutent, SU011248
  Arms: A
Drug: mFOLFOX6 — FOLFOX will be administered every 2 weeks, using the modified FOLFOX6 (mFOLFOX6) regimen, consisting of: - oxaliplatin 85 mg/ m^2 + leucovorin 400 mg/ m^2 (or 200 mg/ m^2 levo-leucovorin) as a 2-hr IV infusion followed by 5-fluorouracil 400 mg/ m^2 IV bolus on day 1 and 5-fluorouracil 2400 mg/ m^2 IV infusion over 46 hours on Days 1 and 2 of each 2 week cycle
  Arms: A
Drug: bevacizumab — Bevacizumab: 5 mg/kg, IV infusion, every 2 weeks.
  Other Names: Avastin
  Arms: B
Drug: mFOLFOX6 — FOLFOX will be administered every 2 weeks, using the modified FOLFOX6 (mFOLFOX6) regimen, consisting of: - oxaliplatin 85 mg/ m^2 + leucovorin 400 mg/ m^2 (or 200 mg/ m^2 levo-leucovorin) as a 2-hr IV infusion followed by 5-fluorouracil 400 mg/ m^2 IV bolus on day 1 and 5-fluorouracil 2400 mg/ m^2 IV infusion over 46 hours on Days 1 and 2 of each 2 week cycle
  Arms: B

SUMMARY:
This study will compare the safety and efficacy of sunitinib in combination with FOLFOX versus bevacizumab in combination with FOLFOX for the treatment of patients with metastatic colorectal cancer who have not been treated before.

DETAILED DESCRIPTION:
The study was terminated on April 26, 2010 due to lack of efficacy, as determined during the interim analysis of data in April 2010, showing that the study did not meet its primary endpoint to demonstrate a statistically significant improvement in PFS. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the colon or rectum with locally advanced or metastatic disease
* Evidence of measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST)
* Eastern Cooperative Oncology Group (ECOG) 0 or 1

Exclusion Criteria:

* Previous treatment with Sutent, Avastin, or any other systemic therapy for locally advanced or metastatic colorectal cancer
* Less than 6 months since completion of adjuvant chemotherapy to documentation of recurrent disease
* History of cardiac disease
* Brain mets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2008-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (84):
- United States (68):
  - Pfizer Investigational Site, Fairhope, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Bentonville, Arkansas
  - Pfizer Investigational Site, Fayetteville, Arkansas
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Bakersfield, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Lancaster, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Mission Hills, California
  - Pfizer Investigational Site, Northrige, California
  - Pfizer Investigational Site, Oxnard, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Redondo Beach, California
  - Pfizer Investigational Site, Santa Barbara, California
  - Pfizer Investigational Site, Santa Maria, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Solvang, California
  - Pfizer Investigational Site, Valencia, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jacksonville Beach, Florida
  - Pfizer Investigational Site, Jasonville, Florida
  - Pfizer Investigational Site, Orange Park, Florida
  - Pfizer Investigational Site, Palatka, Florida
  - Pfizer Investigational Site, Saint Augustine, Florida
  - Pfizer Investigational Site, Stuart, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Sandy Springs, Georgia
  - Pfizer Investigational Site, Maryville, Illinois
  - Pfizer Investigational Site, Chanute, Kansas
  - Pfizer Investigational Site, Dodge City, Kansas
  - Pfizer Investigational Site, El Dorado, Kansas
  - Pfizer Investigational Site, Independence, Kansas
  - Pfizer Investigational Site, Kingman, Kansas
  - Pfizer Investigational Site, Liberal, Kansas
  - Pfizer Investigational Site, Newton, Kansas
  - Pfizer Investigational Site, Parsons, Kansas
  - Pfizer Investigational Site, Salina, Kansas
  - Pfizer Investigational Site, Wellington, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Winfield, Kansas
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Columbus, Mississippi
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Meadowbrook, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Radnor, Pennsylvania
  - Pfizer Investigational Site, Willow Grove, Pennsylvania
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Lubbock, Texas
  - Pfizer Investigational Site, Wenatchee, Washington
- Denmark (3):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Herlev
  - Pfizer Investigational Site, Koebenhavn OE
- Germany (7):
  - Pfizer Investigational Site, Aschaffenburg
  - Pfizer Investigational Site, Bad Saarow
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Düsseldorf
  - Pfizer Investigational Site, Magdeburg
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Regensburg
- Japan (6):
  - Pfizer Investigational Site, Kashiwa, Chiba
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Kitaadachi-gun, Ina-cho, Saitama
  - Pfizer Investigational Site, Suntougun, Shizuoka
  - Pfizer Investigational Site, Utsunomiya, Tochigi
  - Pfizer Investigational Site, Chuo-ku, Tokyo

REFERENCES:
- [Derived] Breen DM, Kim H, Bennett D, Calle RA, Collins S, Esquejo RM, He T, Joaquim S, Joyce A, Lambert M, Lin L, Pettersen B, Qiao S, Rossulek M, Weber G, Wu Z, Zhang BB, Birnbaum MJ. GDF-15 Neutralization Alleviates Platinum-Based Chemotherapy-Induced Emesis, Anorexia, and Weight Loss in Mice and Nonhuman Primates. Cell Metab. 2020 Dec 1;32(6):938-950.e6. doi: 10.1016/j.cmet.2020.10.023. Epub 2020 Nov 17. PMID 33207247
- [Derived] Hecht JR, Mitchell EP, Yoshino T, Welslau M, Lin X, Chow Maneval E, Paolini J, Lechuga MJ, Kretzschmar A. 5-Fluorouracil, leucovorin, and oxaliplatin (mFOLFOX6) plus sunitinib or bevacizumab as first-line treatment for metastatic colorectal cancer: a randomized Phase IIb study. Cancer Manag Res. 2015 Jun 15;7:165-73. doi: 10.2147/CMAR.S61408. eCollection 2015. PMID 26109878
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181104&StudyName=Randomized%20Study%20Of%20Sunitinib%20Plus%20FOLFOX%20Versus%20Bevacizumab%20Plus%20FOLFOX%20In%20Metastatic%20Colorectal%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib + mFOLFOX6: Sunitinib 37.5 milligram (mg) capsule daily administered orally in a 4 weeks on, 2 weeks off intermittent dosing regimen along with a modified combination chemotherapy of fluorouracil, lecovorin and oxaliplatin (mFOLFOX6) regimen consisting of oxaliplatin 85 mg per square meter (mg/m^2) and leucovorin 400 mg/m^2 (or levo-leucovorin 200 mg/m^2) as a 2-hour intravenous (IV) infusion followed by an IV bolus of 5-fluorouracil (5-FU) 400 mg/m^2 on Day 1 and 46-hour IV infusion of 5-FU 2,400 mg/m^2 on Days 1 and 2 of each 2 week cycle.
- Bevacizumab + mFOLFOX6: Bevacizumab 5 mg/kilogram (mg/kg) administered as 90 minute IV infusion every 2 weeks along with mFOLFOX6 regimen consisting of oxaliplatin 85 mg/m^2 and leucovorin 400 mg/m^2 (or levo-leucovorin 200 mg/m^2) as a 2-hour IV infusion followed by an IV bolus of 5-FU 400 mg/m^2 on Day 1 and a 46-hour IV infusion of 5-FU 2,400 mg/m^2 on Days 1 and 2 of each 2 week cycle.
Period: Overall Study
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Started | 96 | 95
Completed | 0 | 0
Not Completed | 96 | 95
Not completed — Adverse Event | 14 | 10
Not completed — Withdrawal by Subject | 4 | 20
Not completed — Death | 1 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Objective progression or relapse | 47 | 41
Not completed — Study terminated by sponsor | 16 | 3
Not completed — Other | 7 | 14
Not completed — Global deterioration of health status | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib + mFOLFOX6: Sunitinib 37.5 mg capsule daily administered orally in a 4 weeks on, 2 weeks off intermittent dosing regimen along with a modified combination chemotherapy of fluorouracil, leucovorin and oxaliplatin (mFOLFOX6) regimen consisting of oxaliplatin 85 mg/m^2 and leucovorin 400 mg/m^2 (or levo-leucovorin 200 mg/m^2) as a 2-hour IV infusion followed by an IV bolus of 5-FU 400 mg/m^2 on Day 1 and 46-hour IV infusion of 5-FU 2,400 mg/m^2 on Days 1 and 2 of each 2 week cycle.
- Bevacizumab + mFOLFOX6: Bevacizumab 5 mg/kg administered as 90 minute IV infusion every 2 weeks along with mFOLFOX6 regimen consisting of oxaliplatin 85 mg/m^2 and leucovorin 400 mg/m^2 (or levo-leucovorin 200 mg/m^2) as a 2-hour IV infusion followed by an IV bolus of 5-FU 400 mg/m^2 on Day 1 and 46-hour IV infusion of 5-FU 2,400 mg/m^2 on Days 1 and 2 of each 2 week cycle.
- Total: Total of all reporting groups
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6 | Total
Number analyzed (Participants) | 96 | 95 | 191
Age Continuous [Mean (Standard Deviation); unit: Years] | 60.60 (9.26) | 59.10 (10.81) | 59.90 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 33 | 68
  Male | 61 | 62 | 123

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline, at every 8-week intervals for 18 months then every 12 weeks thereafter until disease progression (up to Week 115)
Population: The Full Analysis (FA) set included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug according to the randomization schedule, or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 96 | 95
Weeks | 40.50 [39.50 to 44.20] | 67.00 [41.60 to 67.00]
Statistical Analysis 1: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; P-value was calculated from a 1-sided, log-rank test stratified for Eastern Cooperative Oncology Group (ECOG) Performance Status (0 vs. 1), Baseline Lactate Dehydrogenase (LDH): greater than (>) 1.5 vs. less than or equal to (<=) 1.5 * upper limit of normal range (ULN), and Prior Adjuvant Treatment (yes vs. no); Test type: Superiority or Other; p = 0.9963, Log Rank; Hazard Ratio (HR) = 2.705, 95% CI 2-sided [1.272 to 5.751]

2. Secondary Outcome: Overall Survival (OS)
Description: Time in weeks from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 7. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline, at every 8-week intervals for 18 months, and then every 12 weeks thereafter up to every 2 months until death (up to Week 115)
Population: The FA set included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug according to the randomization schedule, or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 96 | 95
Weeks | 84.30 [84.30 to NA] — Upper limit of the confidence interval (C.I) was not reachable as data was not matured at the time of the analysis. | NA [NA to NA] — Median OS could not be determined as data was not matured at the time of the analysis.
Statistical Analysis 1: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; P-value was calculated from a 1-sided, log-rank test stratified for ECOG Performance Status (0 vs. 1), Baseline LDH: >1.5 vs. <=1.5 * ULN, and Prior Adjuvant Treatment (yes vs. no); Test type: Superiority or Other; p = 0.9289, Log Rank; Hazard Ratio (HR) = 1.618, 95% CI 2-sided [0.845 to 3.096]

3. Secondary Outcome: One Year Survival Probability
Description: One year survival probability was defined as the probability of survival at one year after the first dose of study treatment.
Time Frame: Baseline, at every 8-week intervals for 18 months, and then every 12 weeks thereafter up to every 2 months until death (up to 1 year)
Population: Data was not analyzed due to early study termination.
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Two Year Survival Probability
Description: Two year survival probability was defined as the probability of survival at two years after the first dose of study treatment.
Time Frame: Baseline, at every 8-week intervals for 18 months, and then every 12 weeks thereafter up to every 2 months until death (up to 2 years)
Population: Data was not analyzed due to early study termination.
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed response were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as disappearance of all lesions (target and/or non target). PR were those with at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent.
Time Frame: Baseline until disease progression or discontinuation of the study, at every 8-week intervals for 18 months, and then every 12 weeks thereafter up to Week 115
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 96 | 95
Percentage of participants | 41.70 [33.56 to 54.75] | 37.90 [29.81 to 50.87]
Statistical Analysis 1: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Test type: Superiority or Other; p = 0.5898, Chi-squared; F-Distribution = 3.956, 95% CI 2-sided [-10.412 to 18.324]

6. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 5
Population: Data was not analyzed due to early study termination.
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Treatment - Colorectal (FACT-C) Score
Description: FACT-C used for assessment of health-related quality of life (QoL) in participants with cancer. It consists of 36 items, summarized to 5 subscales:physical well-being (PWB) (7 items), functional well-being (FWB) (7 items), social/family well-being (SWB) (7 items); all 3 subscales range from 0 to 28, emotional well-being (EWB) (6 items) range from 0 to 24, colorectal cancer subscale (9 items) range from 0 to 36; higher subscale score=better QoL. All single-item measures range from 0='Not at all' to 4='Very much'. Total possible score range: 0 to 144. High scale score represents a better QoL.
Time Frame: Baseline [Day (D) 1 of Cycle (C) 1] then every 3 cycles thereafter and at the end of treatment (EOT) or withdrawal visit (up to Week 115)
Population: FA set included participants randomized with study drug assignment, regardless of whether participants received study drug, or received a different drug from that to which they were randomized. Here "n" signifies those participants evaluated for this measure at specific time point for each cohort respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 96 | 95
Units on a scale
  PWB Baseline (n= 93, 90) | 23.21 (4.108) | 23.29 (4.324)
  PWB Change at C4 D1 (n=80, 82) | -2.65 (4.132) | -1.24 (4.930)
  PWB Change at C7 D1 (n=59, 75) | -3.39 (5.532) | -1.94 (4.217)
  PWB Change at C10 D1 (n=45, 62) | -3.66 (4.732) | -1.85 (4.690)
  PWB Change at C13 D1 (n=34, 40) | -3.88 (4.969) | -2.24 (4.364)
  PWB Change at C16 D1 (n=25, 32) | -3.88 (4.850) | -2.83 (4.937)
  PWB Change at C19 D1 (n=13, 23) | -3.46 (4.977) | -1.49 (4.308)
  PWB Change at C22 D1 (n=6, 20) | -1.67 (4.885) | -2.08 (3.429)
  PWB Change at C25 D1 (n=1, 15) | 7.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -1.90 (3.762)
  PWB Change at C28 D1 (n=1, 10) | 4.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -1.6 (5.15)
  PWB Change at C31 D1 (n=1, 4) | 3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -2.8 (6.18)
  PWB Change at C34 D1 (n=1, 1) | 6.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  PWB Change at C37 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  PWB Change at C40 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  PWB Change at C43 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  PWB Change at C46 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  PWB Change at C49 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  PWB Change at EOT (n=57, 43) | -4.16 (4.686) | -3.52 (6.222)
  SWB Baseline (n=93, 88) | 23.42 (4.679) | 23.16 (4.442)
  SWB Change at C4 D1 (n=80, 81) | 0.03 (3.129) | 0.31 (3.823)
  SWB Change at C7 D1 (n=59, 73) | -0.24 (3.941) | 0.27 (3.931)
  SWB Change at C10 D1 (n=45, 60) | -0.89 (3.781) | 0.05 (3.753)
  SWB Change at C13 D1 (n=34, 39) | -0.24 (2.486) | -1.33 (4.278)
  SWB Change at C16 D1 (n=25, 31) | -0.64 (3.369) | -1.24 (4.415)
  SWB Change at C19 D1 (n=13, 23) | -0.79 (2.024) | -1.47 (4.751)
  SWB Change at C22 D1 (n=6, 20) | -0.67 (2.065) | -1.18 (3.787)
  SWB Change at C25 D1 (n=1, 15) | -4.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -0.06 (4.191)
  SWB Change at C28 D1 (n=1, 10) | -3.50 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -0.65 (4.627)
  SWB Change at C31 D1 (n=1, 4) | -4.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 3.58 (3.233)
  SWB Change at C34 D1 (n=1, 1) | -3.50 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 1.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  SWB Change at C37 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  SWB Change at C 40 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  SWB Change at C43 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  SWB Change at C46 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  SWB Change at C49 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  SWB Change at EOT (n=57, 43) | -0.35 (3.501) | -0.63 (2.902)
  EWB Baseline (n=93, 90) | 16.74 (4.342) | 17.30 (3.995)
  EWB Change at C4 D1 (n=80, 82) | 0.95 (3.505) | 1.40 (4.108)
  EWB Change at C7 D1 (n=59, 75) | 1.65 (3.108) | 1.71 (4.036)
  EWB Change at C10 D1 (n=45, 62) | 1.40 (4.014) | 1.65 (4.121)
  EWB Change at C13 D1 (n=34, 40) | 1.3 (4.45) | 1.4 (4.30)
  EWB Change at C16 D1 (n=25, 32) | 0.84 (3.934) | 0.96 (4.511)
  EWB Change at C19 D1 (n=13, 23) | 1.2 (2.92) | 1.8 (4.56)
  EWB Change at C22 D1 (n=6, 20) | 0.2 (3.66) | 1.1 (3.39)
  EWB Change at C25 D1 (n=1, 15) | 4.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -0.3 (5.32)
  EWB Change at C28 D1 (n=1, 10) | 4.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.1 (3.45)
  EWB Change at C31 D1 (n=1, 4) | 2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.3 (4.50)
  EWB Change at C34 D1 (n=1, 1) | 4.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  EWB Change at C37 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  EWB Change at C40 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  EWB Change at C43 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  EWB Change at C46 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  EWB Change at C49 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  EWB Change at EOT (n=57, 43) | 0.35 (4.805) | 0.77 (4.942)
  FWB Baseline (n=93, 89) | 17.88 (5.818) | 17.29 (6.328)
  FWB Change at C4 D1 (n=80, 81) | -0.78 (5.007) | 1.56 (5.536)
  FWB Change at C7 D1 (n=59, 74) | -0.02 (5.425) | 1.02 (5.493)
  FWB Change at C10 D1 (n=45, 61) | -0.35 (4.471) | 0.74 (5.884)
  FWB Change at C13 D1 (n=34, 40) | -0.4 (5.02) | 0.8 (5.88)
  FWB Change at C16 D1 (n=24, 31) | -0.7 (3.65) | -0.7 (4.95)
  FWB Change at C19 D1 (n=13, 22) | -0.3 (3.88) | 0.1 (6.11)
  FWB Change at C22 D1 (n=6, 19) | 0.7 (6.35) | -0.8 (4.72)
  FWB Change at C25 D1 (n=1, 14) | 12.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -1.0 (4.40)
  FWB Change at C28 D1 (n=1, 9) | 13.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -0.8 (4.74)
  FWB Change at C31 D1 (n=1, 3) | 6.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 1.0 (3.61)
  FWB Change at C34 D1 (n=1, 1) | 12.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  FWB Change at C37 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  FWB Change at C40 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  FWB Change at C43 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  FWB Change at C46 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  FWB Change at C49 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -3.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  FWB Change at EOT (n=56, 43) | 1.62 (5.394) | 0.14 (6.075)
  CCS Baseline (n=93, 90) | 20.93 (4.733) | 21.26 (5.064)
  CCS Change at C4 D1 (n=78, 82) | -1.49 (4.228) | -0.13 (4.485)
  CCS Change at C7 D1 (n=60, 75) | -1.00 (5.193) | -0.26 (4.726)
  CCS Change at C10 D1 (n=45, 62) | -1.03 (4.859) | -0.16 (5.474)
  CCS Change at C13 D1 (n=34, 40) | -1.33 (5.224) | -0.20 (5.105)
  CCS Change at C16 D1 (n=25, 32) | -1.32 (4.425) | -1.25 (5.086)
  CCS Change at C19 D1 (n=13, 23) | -2.13 (4.732) | -0.36 (4.754)
  CCS Change at C22 D1 (n=6, 20) | -0.92 (5.219) | 0.15 (3.815)
  CCS Change at C25 D1 (n=1, 15) | 1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 1.3 (5.55)
  CCS Change at C28 D1 (n=1, 10) | -2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.4 (5.46)
  CCS Change at C31 D1 (n=1, 4) | -2.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 1.8 (4.35)
  CCS Change at C34 D1 (n=1, 1) | -1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  CCS Change at C37 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  CCS Change at C40 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  CCS Change at C43 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -1.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  CCS Change at C46 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  CCS Change at C49 D1 (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  CCS Change at EOT (n=55, 43) | -1.06 (4.942) | -0.48 (5.679)
Statistical Analysis 1: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C4 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.0515, t-test, 2 sided; Mean Difference (Net) = -1.40, 95% CI 2-sided [-2.82 to 0.01]
Statistical Analysis 2: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C7 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.0876, t-test, 2 sided; Mean Difference (Net) = -1.45, 95% CI 2-sided [-3.11 to 0.22]
Statistical Analysis 3: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C10 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.0522, t-test, 2 sided; Mean Difference (Net) = -1.81, 95% CI 2-sided [-3.64 to 0.02]
Statistical Analysis 4: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C13 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.1339, t-test, 2 sided; Mean Difference (Net) = -1.64, 95% CI 2-sided [-3.81 to 0.52]
Statistical Analysis 5: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C16 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.4233, t-test, 2 sided; Mean Difference (Net) = -1.05, 95% CI 2-sided [-3.68 to 1.57]
Statistical Analysis 6: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C19 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.2211, t-test, 2 sided; Mean Difference (Net) = -1.97, 95% CI 2-sided [-5.18 to 1.24]
Statistical Analysis 7: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C22 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.8184, t-test, 2 sided; Mean Difference (Net) = 0.41, 95% CI 2-sided [-3.22 to 4.04]
Statistical Analysis 8: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C25 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.0380, t-test, 2 sided; Mean Difference (Net) = 8.90, 95% CI 2-sided [0.57 to 17.23]
Statistical Analysis 9: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C28 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.3266, t-test, 2 sided; Mean Difference (Net) = 5.60, 95% CI 2-sided [-6.61 to 17.81]
Statistical Analysis 10: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C31 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.4667, t-test, 2 sided; Mean Difference (Net) = 5.75, 95% CI 2-sided [-16.26 to 27.76]
Statistical Analysis 11: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (C34 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 12: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in PWB between treatment arms (EOT) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.5587, t-test, 2 sided; Mean Difference (Net) = -0.64, 95% CI 2-sided [-2.80 to 1.52]
Statistical Analysis 13: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C4 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.6122, t-test, 2 sided; Mean Difference (Net) = -0.28, 95% CI 2-sided [-1.37 to 0.81]
Statistical Analysis 14: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C7 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.4642, t-test, 2 sided; Mean Difference (Net) = -0.51, 95% CI 2-sided [-1.87 to 0.86]
Statistical Analysis 15: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C10 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.2105, t-test, 2 sided; Mean Difference (Net) = -0.94, 95% CI 2-sided [-2.41 to 0.54]
Statistical Analysis 16: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C13 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.1950, t-test, 2 sided; Mean Difference (Net) = 1.09, 95% CI 2-sided [-0.57 to 2.76]
Statistical Analysis 17: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C16 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.5779, t-test, 2 sided; Mean Difference (Net) = 0.60, 95% CI 2-sided [-1.55 to 2.75]
Statistical Analysis 18: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C19 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.6314, t-test, 2 sided; Mean Difference (Net) = 0.67, 95% CI 2-sided [-2.15 to 3.50]
Statistical Analysis 19: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C22 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.7554, t-test, 2 sided; Mean Difference (Net) = 0.51, 95% CI 2-sided [-2.85 to 3.87]
Statistical Analysis 20: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C25 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.3781, t-test, 2 sided; Mean Difference (Net) = -3.94, 95% CI 2-sided [-13.22 to 5.34]
Statistical Analysis 21: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C28 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.5715, t-test, 2 sided; Mean Difference (Net) = -2.85, 95% CI 2-sided [-13.83 to 8.13]
Statistical Analysis 22: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C31 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.1271, t-test, 2 sided; Mean Difference (Net) = -7.58, 95% CI 2-sided [-19.08 to 3.93]
Statistical Analysis 23: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (C34 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 24: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in SWB between treatment arms (EOT) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.6785, t-test, 2 sided; Mean Difference (Net) = 0.27, 95% CI 2-sided [-1.03 to 1.58]
Statistical Analysis 25: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C4 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.4623, t-test, 2 sided; Mean Difference (Net) = -0.44, 95% CI 2-sided [-1.63 to 0.74]
Statistical Analysis 26: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C7 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.9302, t-test, 2 sided; Mean Difference (Net) = -0.06, 95% CI 2-sided [-1.31 to 1.20]
Statistical Analysis 27: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C10 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.7502, t-test, 2 sided; Mean Difference (Net) = -0.25, 95% CI 2-sided [-1.84 to 1.33]
Statistical Analysis 28: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C13 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.9335, t-test, 2 sided; Mean Difference (Net) = -0.09, 95% CI 2-sided [-2.12 to 1.95]
Statistical Analysis 29: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C16 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.9191, t-test, 2 sided; Mean Difference (Net) = -0.12, 95% CI 2-sided [-2.40 to 2.17]
Statistical Analysis 30: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C19 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.6750, t-test, 2 sided; Mean Difference (Net) = -0.60, 95% CI 2-sided [-3.46 to 2.27]
Statistical Analysis 31: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C22 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.5874, t-test, 2 sided; Mean Difference (Net) = -0.88, 95% CI 2-sided [-4.20 to 2.43]
Statistical Analysis 32: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C25 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.4507, t-test, 2 sided; Mean Difference (Net) = 4.27, 95% CI 2-sided [-7.53 to 16.06]
Statistical Analysis 33: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C28 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.3087, t-test, 2 sided; Mean Difference (Net) = 3.90, 95% CI 2-sided [-4.28 to 12.08]
Statistical Analysis 34: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C31 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.9635, t-test, 2 sided; Mean Difference (Net) = -0.25, 95% CI 2-sided [-16.26 to 15.76]
Statistical Analysis 35: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (C34 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 36: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in EWB between treatment arms (EOT) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.6699, t-test, 2 sided; Mean Difference (Net) = -0.42, 95% CI 2-sided [-2.37 to 1.53]
Statistical Analysis 37: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C4 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.0055, t-test, 2 sided; Mean Difference (Net) = -2.34, 95% CI 2-sided [-3.98 to -0.70]
Statistical Analysis 38: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C7 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.2793, t-test, 2 sided; Mean Difference (Net) = -1.04, 95% CI 2-sided [-2.92 to 0.85]
Statistical Analysis 39: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C10 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.2999, t-test, 2 sided; Mean Difference (Net) = -1.09, 95% CI 2-sided [-3.17 to 0.99]
Statistical Analysis 40: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C13 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.3270, t-test, 2 sided; Mean Difference (Net) = -1.27, 95% CI 2-sided [-3.82 to 1.29]
Statistical Analysis 41: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C16 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.9779, t-test, 2 sided; Mean Difference (Net) = 0.03, 95% CI 2-sided [-2.39 to 2.45]
Statistical Analysis 42: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C19 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.8344, t-test, 2 sided; Mean Difference (Net) = -0.40, 95% CI 2-sided [-4.25 to 3.45]
Statistical Analysis 43: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C22 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.5494, t-test, 2 sided; Mean Difference (Net) = 1.46, 95% CI 2-sided [-3.50 to 6.41]
Statistical Analysis 44: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C25 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.0136, t-test, 2 sided; Mean Difference (Net) = 13.00, 95% CI 2-sided [3.15 to 22.85]
Statistical Analysis 45: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C28 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.0247, t-test, 2 sided; Mean Difference (Net) = 13.78, 95% CI 2-sided [2.26 to 25.29]
Statistical Analysis 46: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C31 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.3527, t-test, 2 sided; Mean Difference (Net) = 5.00, 95% CI 2-sided [-12.91 to 22.91]
Statistical Analysis 47: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (C34 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 48: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in FWB between treatment arms (EOT) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.1309, t-test, 2 sided; Mean Difference (Net) = -1.76, 95% CI 2-sided [-4.05 to 0.53]
Statistical Analysis 49: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C4 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.0510, t-test, 2 sided; Mean Difference (Net) = -1.36, 95% CI 2-sided [-2.72 to 0.01]
Statistical Analysis 50: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C7 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.3858, t-test, 2 sided; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-2.44 to 0.95]
Statistical Analysis 51: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C10 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.3943, t-test, 2 sided; Mean Difference (Net) = -0.88, 95% CI 2-sided [-2.90 to 1.15]
Statistical Analysis 52: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C13 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.3499, t-test, 2 sided; Mean Difference (Net) = -1.13, 95% CI 2-sided [-3.53 to 1.27]
Statistical Analysis 53: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C16 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.9567, t-test, 2 sided; Mean Difference (Net) = -0.07, 95% CI 2-sided [-2.64 to 2.50]
Statistical Analysis 54: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C19 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.2901, t-test, 2 sided; Mean Difference (Net) = -1.77, 95% CI 2-sided [-5.12 to 1.58]
Statistical Analysis 55: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C22 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.5857, t-test, 2 sided; Mean Difference (Net) = -1.07, 95% CI 2-sided [-5.05 to 2.92]
Statistical Analysis 56: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C25 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.9635, t-test, 2 sided; Mean Difference (Net) = -0.27, 95% CI 2-sided [-12.56 to 12.02]
Statistical Analysis 57: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C28 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.6850, t-test, 2 sided; Mean Difference (Net) = -2.40, 95% CI 2-sided [-15.36 to 10.56]
Statistical Analysis 58: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C31 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.4968, t-test, 2 sided; Mean Difference (Net) = -3.75, 95% CI 2-sided [-19.23 to 11.73]
Statistical Analysis 59: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (C34 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 60: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in CCS between treatment arms (EOT) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.5891, t-test, 2 sided; Mean Difference (Net) = -0.58, 95% CI 2-sided [-2.71 to 1.55]

8. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Treatment - Gynecologic Oncology Group Oxaliplatin-Specific Neurotoxicity (FACT&GOG-Ntx) Score
Description: FACT&GOG-Ntx has a 13-item, treatment-specific subscale for patients with neurotoxicity. It is the sum of the PWB (7 items), FWB (7 items), SWB (7 items) and EWB (6 items) subscales plus a 13 item neurotoxicity subscale. Subscale score ranges from 0 to 28 for PWB, FWB, SWB, 0 to 24 for EWB and 0 to 52 for neurotoxicity subscale. Total possible score range is 0 to 160. Higher scores indicates better QoL, fewer disease symptoms, and/or fewer side effects of treatment and lower scores indicate worse QoL and a greater impact of disease symptoms and/or side effects.
Time Frame: Baseline (D1 of C1) then every 3 cycles thereafter and at the EOT or withdrawal visit (up to 115 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Number analyzed (Participants) | 96 | 95
Units on a scale
  Baseline (Neurotoxicity) (n=90, 93) | 44.04 (4.853) | 44.41 (4.808)
  Change at C4 D1 (Neurotoxicity) (n=75, 80) | -4.73 (6.270) | -4.10 (5.514)
  Change at C7 D1 (Neurotoxicity) (n=60, 74) | -6.20 (7.504) | -5.76 (5.560)
  Change at C10 D1 (Neurotoxicity) (n=45, 61) | -10.21 (8.800) | -7.45 (7.231)
  Change at C13 D1 (Neurotoxicity) (n=34, 40) | -13.96 (9.494) | -12.73 (9.420)
  Change at C16 D1 (Neurotoxicity) (n=24, 31) | -15.58 (8.356) | -14.55 (10.977)
  Change at C19 D1 (Neurotoxicity) (n=13, 23) | -12.4 (8.58) | -16.6 (9.71)
  Change at C22 D1 (Neurotoxicity) (n=5, 20) | -5.60 (6.914) | -13.87 (8.122)
  Change at C25 D1 (Neurotoxicity) (n=1, 14) | -13.0 (NA) — Standard deviation was not estimable as only one participant was evaluable. | -16.9 (9.09)
  Change at C28 D1 (Neurotoxicity) (n=1, 10) | -13.0 (NA) — Standard deviation was not estimable as only one participant was evaluable. | -14.0 (8.03)
  Change at C31 D1 (Neurotoxicity) (n=1, 4) | -12.0 (NA) — Standard deviation was not estimable as only one participant was evaluable. | -13.8 (4.11)
  Change at C34 D1 (Neurotoxicity) (n=1, 1) | -12.0 (NA) — Standard deviation was not estimable as only one participant was evaluable. | -9.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at C37 D1 (Neurotoxicity) (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -9.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at C40 D1 (Neurotoxicity) (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -10.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at C43 D1 (Neurotoxicity) (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -10.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at C46 D1 (Neurotoxicity) (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -8.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at C49 D1 (Neurotoxicity) (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -8.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at EOT (Neurotoxicity) (n=56, 43) | -10.71 (9.561) | -9.97 (8.632)
  Baseline (Item 13) (n=90, 93) | 3.8 (0.55) | 3.9 (0.42)
  Change at C4 D1 (Item 13) (n=75, 79) | -0.2 (0.52) | -0.2 (0.65)
  Change at C7 D1 (Item 13) (n=60, 74) | -0.3 (0.68) | -0.2 (0.56)
  Change at C10 D1 (Item 13) (n=45, 61) | -0.4 (0.87) | -0.2 (0.79)
  Change at C13 D1 (Item 13) (n=34, 40) | -0.4 (0.86) | -0.2 (0.68)
  Change at C16 D1 (Item 13) (n=24, 31) | -0.6 (1.03) | -0.6 (0.89)
  Change at C19 D1 (Item 13) (n=13, 23) | -0.3 (0.48) | -0.7 (1.19)
  Change at C22 D1 (Item 13) (n=5, 20) | -0.4 (0.55) | -0.4 (0.88)
  Change at C25 D1 (Item 13) (n=1, 14) | 0.0 (NA) — Standard deviation was not estimable as only one participant was evaluable. | -0.6 (0.94)
  Change at C28 D1 (Item 13) (n=1, 10) | -1.0 (NA) — Standard deviation was not estimable as only one participant was evaluable. | -0.6 (1.07)
  Change at C31 D1 (Item 13) (n=1, 4) | 0.0 (NA) — Standard deviation was not estimable as only one participant was evaluable. | -1.3 (0.96)
  Change at C34 D1 (Item 13) (n=1, 1) | -1.0 (NA) — Standard deviation was not estimable as only one participant was evaluable. | -1.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at C37 D1 (Item 13) (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | -1.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at C40 D1 (Item 13) (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at C43 D1 (Item 13) (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at C46 D1 (Item 13) (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at C49 D1 (Item 13) (n=0, 1) | NA (NA) — Data was not analyzed due to early study termination. | 0.0 (NA) — Standard deviation was not estimable as only one participant was evaluable.
  Change at EOT (Item 13) (n=56, 43) | -0.4 (0.85) | -0.3 (0.78)
Statistical Analysis 1: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C4 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.5081, t-test, 2 sided; Mean Difference (Net) = -0.63, 95% CI 2-sided [-2.50 to 1.24]
Statistical Analysis 2: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C7 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.6977, t-test, 2 sided; Mean Difference (Net) = -0.44, 95% CI 2-sided [-2.67 to 1.79]
Statistical Analysis 3: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C10 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.0797, t-test, 2 sided; Mean Difference (Net) = -2.76, 95% CI 2-sided [-5.85 to 0.33]
Statistical Analysis 4: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C13 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.5808, t-test, 2 sided; Mean Difference (Net) = -1.22, 95% CI 2-sided [-5.62 to 3.17]
Statistical Analysis 5: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C16 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.7046, t-test, 2 sided; Mean Difference (Net) = -1.03, 95% CI 2-sided [-6.44 to 4.38]
Statistical Analysis 6: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C19 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.2052, t-test, 2 sided; Mean Difference (Net) = 4.18, 95% CI 2-sided [-2.40 to 10.76]
Statistical Analysis 7: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C22 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.0483, t-test, 2 sided; Mean Difference (Net) = 8.27, 95% CI 2-sided [0.07 to 16.46]
Statistical Analysis 8: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C25 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.6832, t-test, 2 sided; Mean Difference (Net) = 3.93, 95% CI 2-sided [-16.41 to 24.26]
Statistical Analysis 9: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C28 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.9081, t-test, 2 sided; Mean Difference (Net) = 1.00, 95% CI 2-sided [-18.05 to 20.05]
Statistical Analysis 10: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C31 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.7289, t-test, 2 sided; Mean Difference (Net) = 1.75, 95% CI 2-sided [-12.88 to 16.38]
Statistical Analysis 11: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (C34 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 12: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in neurotoxicity between treatment arms (EOT) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.6921, t-test, 2 sided; Mean Difference (Net) = -0.74, 95% CI 2-sided [-4.43 to 2.95]
Statistical Analysis 13: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C4 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.9788, t-test, 2 sided; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.19 to 0.19]
Statistical Analysis 14: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C7 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.2747, t-test, 2 sided; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.33 to 0.09]
Statistical Analysis 15: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C10 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.2776, t-test, 2 sided; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.50 to 0.14]
Statistical Analysis 16: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C13 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.1403, t-test, 2 sided; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.62 to 0.09]
Statistical Analysis 17: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C16 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.9151, t-test, 2 sided; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.55 to 0.50]
Statistical Analysis 18: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C19 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.3277, t-test, 2 sided; Mean Difference (Net) = 0.34, 95% CI 2-sided [-0.36 to 1.05]
Statistical Analysis 19: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C22 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 1.0000, t-test, 2 sided; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.86 to 0.86]
Statistical Analysis 20: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C25 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.5661, t-test, 2 sided; Mean Difference (Net) = 0.57, 95% CI 2-sided [-1.53 to 2.67]
Statistical Analysis 21: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C28 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.7309, t-test, 2 sided; Mean Difference (Net) = -0.40, 95% CI 2-sided [-2.95 to 2.15]
Statistical Analysis 22: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C31 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.3273, t-test, 2 sided; Mean Difference (Net) = 1.25, 95% CI 2-sided [-2.16 to 4.66]
Statistical Analysis 23: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (C34 of D1) was analyzed from a two-sample t-test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [0 to 0]
Statistical Analysis 24: Comparison: Sunitinib + mFOLFOX6 vs Bevacizumab + mFOLFOX6; Differences in item 13 between treatment arms (EOT) was analyzed from a two-sample t-test; Test type: Superiority or Other; p = 0.7108, t-test, 2 sided; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.39 to 0.27]

ADVERSE EVENTS:
Description: Same event may appear as both AE and SAE. But distinct events are presented. Event may be serious in 1 subject and nonserious in another, or 1 subject may have both serious, nonserious event. At risk population=participants with metastatic colorectal cancer, with at least 1 dose of study medication; Sunitinib+mFOLFOX6=96, Bevacizumab+mFOLFOX6=93.
Arm/Group | Sunitinib + mFOLFOX6 | Bevacizumab + mFOLFOX6
Serious Adverse Events (participants affected / at risk) | 36/96 | 30/93
Other Adverse Events (participants affected / at risk) | 96/96 | 93/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + mFOLFOX6 (N=96) | Bevacizumab + mFOLFOX6 (N=93)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Ocular icterus (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Adverse drug reaction (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 2
Device dislocation (General disorders) | 0 | 1
Disease progression (General disorders) | 4 | 3
Medical device complication (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal wall infection (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Haemophilus bacteraemia (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Post procedural infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Hepatectomy (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 3
Haemorrhage (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 2
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + mFOLFOX6 (N=96) | Bevacizumab + mFOLFOX6 (N=93)
Anaemia (Blood and lymphatic system disorders) | 27 | 26
Leukopenia (Blood and lymphatic system disorders) | 21 | 11
Neutropenia (Blood and lymphatic system disorders) | 67 | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 50 | 19
Lacrimation increased (Eye disorders) | 5 | 5
Vision blurred (Eye disorders) | 6 | 3
Abdominal distension (Gastrointestinal disorders) | 6 | 5
Abdominal pain (Gastrointestinal disorders) | 20 | 21
Abdominal pain lower (Gastrointestinal disorders) | 1 | 5
Abdominal pain upper (Gastrointestinal disorders) | 6 | 7
Cheilitis (Gastrointestinal disorders) | 4 | 5
Constipation (Gastrointestinal disorders) | 22 | 30
Diarrhoea (Gastrointestinal disorders) | 66 | 49
Dry mouth (Gastrointestinal disorders) | 11 | 5
Dyspepsia (Gastrointestinal disorders) | 17 | 7
Dysphagia (Gastrointestinal disorders) | 4 | 7
Flatulence (Gastrointestinal disorders) | 5 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 7
Haemorrhoids (Gastrointestinal disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 62 | 57
Oral pain (Gastrointestinal disorders) | 6 | 5
Proctalgia (Gastrointestinal disorders) | 5 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 5
Stomatitis (Gastrointestinal disorders) | 31 | 26
Vomiting (Gastrointestinal disorders) | 33 | 33
Asthenia (General disorders) | 8 | 11
Chest pain (General disorders) | 2 | 10
Chills (General disorders) | 2 | 6
Fatigue (General disorders) | 65 | 62
Mucosal inflammation (General disorders) | 12 | 21
Oedema peripheral (General disorders) | 11 | 5
Pain (General disorders) | 7 | 9
Pyrexia (General disorders) | 21 | 22
Hypersensitivity (Immune system disorders) | 2 | 5
Nasopharyngitis (Infections and infestations) | 4 | 9
Rhinitis (Infections and infestations) | 0 | 7
Upper respiratory tract infection (Infections and infestations) | 4 | 6
Urinary tract infection (Infections and infestations) | 10 | 3
Contusion (Injury, poisoning and procedural complications) | 5 | 1
Blood alkaline phosphatase increased (Investigations) | 5 | 5
Blood potassium decreased (Investigations) | 5 | 1
Haemoglobin decreased (Investigations) | 6 | 2
Neutrophil count decreased (Investigations) | 19 | 8
Platelet count decreased (Investigations) | 17 | 0
Weight decreased (Investigations) | 19 | 16
White blood cell count decreased (Investigations) | 13 | 5
Decreased appetite (Metabolism and nutrition disorders) | 32 | 36
Dehydration (Metabolism and nutrition disorders) | 11 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 10
Dizziness (Nervous system disorders) | 14 | 16
Dysgeusia (Nervous system disorders) | 31 | 21
Headache (Nervous system disorders) | 14 | 22
Hyperaesthesia (Nervous system disorders) | 7 | 8
Hypoaesthesia (Nervous system disorders) | 5 | 5
Neuropathy peripheral (Nervous system disorders) | 39 | 37
Paraesthesia (Nervous system disorders) | 6 | 14
Peripheral sensory neuropathy (Nervous system disorders) | 29 | 33
Polyneuropathy (Nervous system disorders) | 0 | 5
Anxiety (Psychiatric disorders) | 5 | 13
Depression (Psychiatric disorders) | 6 | 11
Insomnia (Psychiatric disorders) | 16 | 20
Proteinuria (Renal and urinary disorders) | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 16
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 30
Hiccups (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 24
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 26 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 9
Rash (Skin and subcutaneous tissue disorders) | 20 | 16
Skin discolouration (Skin and subcutaneous tissue disorders) | 9 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 8
Yellow skin (Skin and subcutaneous tissue disorders) | 9 | 0
Hypertension (Vascular disorders) | 19 | 21
Hypotension (Vascular disorders) | 2 | 6

LIMITATIONS AND CAVEATS:
Due to early study termination, not all data was analyzable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.